CLINICAL TRIAL: NCT07239024
Title: Evaluation of Piezocision Versus Injectable Platelet-rich Fibrin During Orthodontic Canine Retraction: A Comparative Clinical Stud
Brief Title: Evaluation of Piezocision Versus Injectable Platelet-rich Fibrin During Orthodontic Canine Retraction Orthodontic Canine Retraction: A Comparative Clinical Study
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, farouk ahmed hussein, Professor of orthodontics, Al-Azhar University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 1250/5544
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Effect of Piezocision and Injectable Platelets Rich Fibrin on Tooth Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Iprf experimental side (Experimental): Injection of platelet rich fibrin
  Interventions: Procedure: Iprf and piezocision
- iPrf control side (No Intervention)
- Piezocisin experimental side (Experimental): Flapless incision
  Interventions: Procedure: Iprf and piezocision
- Piezocision control sode (No Intervention)

INTERVENTIONS:
Procedure: Iprf and piezocision — Injection of iprf and piezocisin
  Arms: Iprf experimental side; Piezocisin experimental side

SUMMARY:
Comparison of piezocisin and injectable platelets rich fibrin during canine retraction

DETAILED DESCRIPTION:
Evaluation of piezocision versus injectable platelet-rich fibrin during orthodontic canine retraction: A comparative clinical study

ELIGIBILITY:
Inclusion Criteria:. An age ranges from 14-22 years. 2. Crowding or protrusion that require 1st premolars extraction, followed by symmetrical canine retractions.

3. All permanent teeth present, 3rd molars aren't considered. 4. Good oral hygiene. 5. No systemic disease and/or medication that could interfere with orthodontic tooth movement. 6. No previous orthodontic treatment. 7. No evidence of craniofacial anomalies, such as cleft lip and palate or previous history of trauma, bruxism, or parafunction. 8. No tooth size, shape, or root abnormalities visible on patient's radiographic records.

-

Exclusion Criteria:Patients diagnosed to have an indication for non-extraction approach.

2. Poor oral hygiene or periodontally compromised patient.

* 3. Previous orthodontic treatment. 4. Any implanted assistive (e.g., pacemakers, cochlear implants, etc.). 5. Any skeletal dysplasia or craniofacial malformation. 6. Patients with root resorption, impacted canine or dental anomalies. 7. Any systemic diseases or medications that could interfere with orthodontic tooth movement.

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Rate of canine retraction | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- AlAzhar university, Cairo, Egypt